CLINICAL TRIAL: NCT00712777
Title: Relation Between Intraocular Pressure Lowering Effects of Topical Brimonidine and Alpha 2 Receptor Polymorphism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjäger-Mayrl, MD, Department of Clinical Pharmacology
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-230408
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Ocular Physiology; Intraocular Pressure
Keywords: Brimonidine; alpha 2 receptor polymorphism; Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): homozygote mutant: Insertion/Insertion (40 patients)
  Interventions: Drug: Brimonidine 0.2 %
- 2 (Active Comparator): homozygote mutant: Deletion/Deletion (40 patients)
  Interventions: Drug: Brimonidine 0.2 %

INTERVENTIONS:
Drug: Brimonidine 0.2 % — Brimonidine 0.2 % (Alphagan, Irvine, CA, USA), dose: 1 drop per eye

SUMMARY:
Topical brimonidine is a recently introduced alpha 2 receptor agonist which is used in the therapy of intraocular pressure (IOP) reduction in patients with open angle glaucoma. Although adequate IOP reduction is achieved in many patients there is a considerable degree of variability in IOP reduction among subjects. The reason for this interindividual variability is not entirely clear. Obviously differences in pharmacokinetic properties due to variable penetration of the drug through the cornea may be responsible. Alternatively, polymorphisms of the alpha-2 receptor may account for the differences in IOP-lowering efficacy of topical brimonidine. This hypothesis is tested in the present study. Polymorphisms of the alpha-2 receptor have been described in a number of previous studies. In addition, polymorphisms in the alpha-2 receptor gene have been shown to be functionally important, particularly a polymorphism of the alpha-2B receptor, which has a high allele frequency in caucasians.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* IOP between 12 and 16 mmHg
* Normal ophthalmic findings, ametropia < 3 Dpt.
* Results of alpha-2B receptor genotyping; subjects who fall within one of the following groups: group 1: homozygote mutant: I/I (n=40); group 2: homozygote mutant: D/D (n=40)

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | in total 10 minutes
alpha-2B receptor genotyping | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Vienna, Vienna, Austria